CLINICAL TRIAL: NCT05556499
Title: Interactions Between Bone and Parathyroid Tumors in Patiens With Primary Hyperparathyroidism (The PARABONE Study)
Brief Title: The Bone-parathyroid Crosstalk in Primary Hyperparathyroidism
Acronym: PARABONE
Status: Not yet recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: PARABONE (L4126)
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Hyperparathyroidism, Primary; Osteoporosis; Parathyroid Neoplasms
MeSH Terms: conditions — Hyperparathyroidism, Primary; Osteoporosis; Parathyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Parathyroid tumor samples derived from patients undergoing excisional surgery and peripheral blood samples at diagnosis will be collected
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HPT patients: Patients with primary hyperparathyroidism at diagnosis (HPT) treated with parathyroidectomy (HPT-PTX)
  Interventions: Diagnostic Test: Biomarker assays

INTERVENTIONS:
Diagnostic Test: Biomarker assays — Circulating bone biomarkers assays

SUMMARY:
The PARABONE study aims to investigate the interaction between bone and parathyroid glands in patients with primary hyperparathyroidism (HPT). The study consists of a clinical part aimed at evaluating a series of circulating molecules of bone derivation (osteocalcin, molecules of the WNT pathway, RANKL, osteoprotegerin, Scelrostin, FGF23) in patients with HPT. In particular, the study has as its primary objective to identify the correlation between circulating levels of PTH and levels of GlaOC and GluOC in patients with HPT.

DETAILED DESCRIPTION:
The parathyroid glands are responsible for controlling mineral homeostasis in order to keep circulating calcium levels constant by acting on the target organs, where they induce mobilization of calcium from the bone matrix, and they promote the reabsorption of calcium from the ultra-filtrate at renal level. In turn, kidney and bone can affect the functioning of the parathyroid glands, for example through the action of FGF23 secreted by osteocytes. Primary hyperparathyroidism (HPT) is an endocrine disorder that causes bone demineralization, osteoporosis and fragility fractures, representing a frequent cause of secondary osteoporosis. It is prevalent in postmenopausal women, where it is the third most frequent endocrine pathology after diabetes and thyroid disease. In postmenopausal women, the pattern of demineralization induced by estrogen deficiency may overlap with that secondary to HPT. HPT is sustained by tumors of the parathyroid glands, mainly of a benign nature, associated with inappropriate secretion of parathyroid hormone (PTH), which causes hypercalcemia and bone, kidney and cardiovascular complications. It is known that persistent secondary hyperparathyroidism, such as that induced by idiopathic hypercalciuria or malabsorption related to vitamin D deficiency, can stimulate the proliferation of parathyroid cells and the autonomous hypersecretion of PTH. Therefore, it is conceivable that also alterations in bone metabolism, such as a persistently increased release of osteocalcin (OC), can promote the proliferation of parathyroid cells and/or hypersecretion of PTH. Interestingly, the circulating levels of carboxylated and decarboxylated osteocalcin (GlaOC and GluOC) were found to be increased in patients with HPT. Furthermore, elevated circulating OC levels appear to be predictive of multiglandular disease in HPT patients. Osteoblasts are one of the main targets of PTH action and release biologically active molecules with paracrine and endocrine action, including osteocalcin (GlaOC and GluOC), the molecules of the intracellular signaling pathway WNT and the RANK ligand (Receptor Activator for Nuclear Factor-κB, RANKL). Therefore, it is conceivable that these biologically active molecules released by osteoblasts can induce biological effects of modulating the functioning of parathyroid cells, in a sort of bone-parathyroid regulatory loop, and thus modulate the presentation phenotype and clinical severity of HPT. RANKL and sclerostin are the specific targets of monoclonal anti-osteoporotic treatments currently available; therefore understanding their potential effect on parathyroid function in HPT can provide the rationale for new therapeutic approaches for patients with HPT. The expected results will allow to improve the diagnosis of HPT, in particular to better define the extent of bone compromise related to it, evaluating circulating bone markers so far not explored. The investigators therefore intend to clarify the effect of hormones released by osteoblasts on parathyroid function, taking into account that these hormones are the target of currently available anti-osteoporotic therapies. The translational study will therefore allow to identify new pathogenetic mechanisms in parathyroid tumorigenesis promoted by endocrine factors released by osteoblasts, which will be able to provide potential targets for targeted medical treatments.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the HPT patient group:

* diagnosis of primary hyperparathyroidism according to the most recent guidelines [Marcocci et al. 2015];
* adult patients (age ≥ 18 years);
* signature of the informed consent.

Inclusion criteria for the HPT-PTX patient group:

* diagnosis of primary hyperparathyroidism with indication of surgical removal of the parathyroid tumor according to the most recent guidelines [Marcocci et al. 2015];
* adult patients (age ≥18 years);
* signature of the informed consent.

Exclusion Criteria:

* Criteria for exclusion from the study are:
* age <18 years
* diagnosis of hyperparathyroidism secondary to chronic renal failure or to vitamin D or calcium deficiency;
* pregnancy or breastfeeding (self-declaration)
* lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients aged ≥ 18 years with a diagnosis of HPT according to the most recent guidelines will be enrolled in the study [Marcocci et al. 2015] with and without indication for surgical treatment.
  Serum and plasma samples will be collected from all patients with HPT and parathyroid tumor samples from patients diagnosed with HPT with indication for surgical treatment according to the guidelines [Bilezikian et al. 2014, Marcocci et al. 2015].
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2026-05-24 (Estimated); Study Completion 2026-06-24 (Estimated)

PRIMARY OUTCOMES:
Correlation between circulating GlaOC and PTH levels in HPT patients | 42 months
  The study aims to investigate the effect of the circulating carboxylated osteocalcin isoform (GlaOC) on the biochemical phenotype in patients with HPT

SECONDARY OUTCOMES:
Effects of bone derived molecules on the biochemical phenotypes and parathyroid tumor cells function in HPT patients | 42 months
  Correlation between the clinical and biochemical characteristics of HPT patients with circulating levels of the two isoforms of osteocalcin and other hormones produced by bone (molecules of the WNT pathway, RANKL, Osteoprotegerin, Sclerostin, FGF23, IL-17). Analysis of the expression of circulating lncRNAs and microRNAs in patients with HPT in relation to the osteo-metabolic state. Analysis of the expression pattern of genes involved in parathyroid tumorigenesis and in bone-parathyroid crosstalk, lncRNAs and microRNAs in parathyroid cancer cells in order to further define the heterogeneity of the adenoma histotype in relation to the osteo-metabolic state.Define the biological effect of the hormones released from bone on parathyroid cancer cells. Define the biological effect and the interaction with the parathyroid function of the hormones released from bone in HEK293A models transfected with the CASR and / or transfected with the receptors of the molecules released by bone.

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Corbetta, PhD, MD, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gianotti L, Piovesan A, Croce CG, Pellegrino M, Baffoni C, Cesario F, Visconti G, Borretta G, Tassone F. Interplay between serum osteocalcin and insulin sensitivity in primary hyperparathyroidism. Calcif Tissue Int. 2011 Mar;88(3):231-7. doi: 10.1007/s00223-010-9453-1. Epub 2011 Jan 5. PMID 21207016
- [Result] Marcocci C, Brandi ML, Scillitani A, Corbetta S, Faggiano A, Gianotti L, Migliaccio S, Minisola S. Italian Society of Endocrinology Consensus Statement: definition, evaluation and management of patients with mild primary hyperparathyroidism. J Endocrinol Invest. 2015 May;38(5):577-93. doi: 10.1007/s40618-015-0261-3. Epub 2015 Mar 28. No abstract available. PMID 25820553
- [Result] Maser RE, Lenhard MJ, Pohlig RT, Balagopal PB, Abdel-Misih R. Effect of parathyroidectomy on osteopontin and undercarboxylated osteocalcin in patients with primary hyperparathyroidism. Endocr Res. 2018 Feb;43(1):21-28. doi: 10.1080/07435800.2017.1369432. Epub 2017 Sep 22. PMID 28937873
- [Result] Mendonca ML, Batista SL, Nogueira-Barbosa MH, Salmon CE, Paula FJ. Primary Hyperparathyroidism: The Influence of Bone Marrow Adipose Tissue on Bone Loss and of Osteocalcin on Insulin Resistance. Clinics (Sao Paulo). 2016 Aug;71(8):464-9. doi: 10.6061/clinics/2016(08)09. PMID 27626477
- [Result] Thier M, Daudi S, Bergenfelz A, Almquist M. Predictors of multiglandular disease in primary hyperparathyroidism. Langenbecks Arch Surg. 2018 Feb;403(1):103-109. doi: 10.1007/s00423-017-1647-9. Epub 2018 Jan 2. PMID 29294178
- [Result] Parveen B, Parveen A, Vohora D. Biomarkers of Osteoporosis: An Update. Endocr Metab Immune Disord Drug Targets. 2019;19(7):895-912. doi: 10.2174/1871530319666190204165207. PMID 30727928
- [Result] Bilezikian JP, Brandi ML, Eastell R, Silverberg SJ, Udelsman R, Marcocci C, Potts JT Jr. Guidelines for the management of asymptomatic primary hyperparathyroidism: summary statement from the Fourth International Workshop. J Clin Endocrinol Metab. 2014 Oct;99(10):3561-9. doi: 10.1210/jc.2014-1413. Epub 2014 Aug 27. PMID 25162665